CLINICAL TRIAL: NCT04783675
Title: Efficacy and Safety of Rituximab in the First Episode of Pediatric Idiopathic Nephrotic Syndrome
Acronym: RTXFIRPedINS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Children's Hospital of Nanjing Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Anhui Provincial Children's Hospital (Other); Children's Hospital Affiliated to Zhengzhou University/Henan Children's Hospital (Unknown); The first affiliated hospital of Zhongshan university (Unknown); Shandong Provincial Hospital (Other Government); Xuzhou Children Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTXFIRPedINS
Record Dates: First submitted 2021-02-28; First posted 2021-03-05 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Steroid-Sensitive Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Rituximab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/treatment (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab (375 mg/m2) will be given as a single intravenous infusion after remission

SUMMARY:
The main objective is to demonstrate, from the initial episode of nephrotic syndrome (NS) in children with standard prednisolone treatment, once complete remission has occurred, that the use of Rituximab (a single intravenous infusion of 375 mg/m2) may reduce the risk of subsequent relapse during 12-month of follow-up.

DETAILED DESCRIPTION:
NS is the most frequent glomerular disease in children. Between 80% and 90% of children with steroid-sensitive nephrotic syndrome (SSNS) will relapse following an initial response to corticosteroids. Half of these children will experience frequent relapses (FRNS) or become steroid-dependent (SDNS).

The results of multiple observational studies and randomized control trials have shown that Rituximab, a chimeric monoclonal antibody against the cluster of differentiation antigen 20 (CD20) antigen on B cells, is safe and effective for children with FRNS/SDNS without corticosteroid or immunosuppressive therapy. To the investigators' knowledge, Rituximab has never been investigated for the initial episode of NS with the aim to reduce the subsequent risk of relapse that is a major concern in the management of children with NS.

Children aged 1-18 years with the first episode of the SSNS will be treated with a single intravenous infusion of Rituximab 375 mg/m2. The prednisolone at a dose of 2 mg/kg per day (maximum 60 mg in single or divided doses) for 6 weeks, followed by 1.5 mg/kg (maximum 40 mg) as a single morning dose on alternate days for the next 6 weeks; therapy is then discontinued.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children between 1 and 18 years with Steroid-Sensitive Nephrotic Syndrome
* 2. Estimated glomerular filtration rate (eGFR) ≥90 ml/min per 1.73 m2 at study entry.
* 3. Remission at study entry
* 4.CD20 positive cells in peripheral blood ≥1% total lymphocytes
* 5.No immunosuppressive agents have been used within 3 months of enrollment, except for the use of corticosteroid to treat nephrotic syndrome.
* 6. Provision of consent by a legal representative (parents or legal guardians) using a document approved by the institutional review board after receiving an adequate explanation regarding the implementation of this clinical trial. For children/youth ages 10-18, written assent is required using age-appropriate and background-appropriate documents.

Exclusion Criteria:

* 1.Diagnosis of secondary NS
* 2.Patients showing one of the following abnormal clinical laboratory values: leukopenia (white blood cell count ≤3.0*109/L); moderate and severe anemia (hemoglobin <9.0g/dL); thrombocytopenia (platelet count <100*1012/ L); positivity of autoimmunity tests (ANA, Anti DNA antibody, ANCA) or reduced C3 levels; Positive for hepatitis B surface (HBs) antigen, HBs antibody, hepatitis B core (HBc) antibody, or hepatitis C virus (HCV) antibody ; Positive for HIV antibody; Alanine aminotransferase (ALT) > 2.5× upper limit of normal value. Aspartate aminotransferase (AST) > 2.5× upper limit of normal value.
* 3. Presence or history of severe or opportunistic infections within 6 months before assignment; Presence of active tuberculosis or with a history of tuberculosis or in whom tuberculosis is suspected; Presence or history of chronic active infections such as Epstein-Barr virus and CMV virus; presence or history of active hepatitis B or hepatitis C or hepatitis B virus carrier. Presence of human immunodeficiency virus (HIV) infection or other active viral infections
* 4. Receipt of a live vaccine within 4 weeks before enrollment.
* 5. Prior receipt of monoclonal antibodies of any type
* 6. History of angina pectoris, cardiac failure, myocardial infarction, or serious arrhythmia，or poorly controlled hypertension
* 7. Presence or history of autoimmune diseases or vascular purpura.
* 8. Presence or history of malignant tumor
* 9. History of organ transplantation (excluding corneal and hair transplants).
* 10. Patients with a known allergy to steroid and their excipients or to Rituximab and its excipients or to acetaminophen and its excipients or to cetirizine and its excipients or to the protein of murine origin
* 11. Assessed to be unfit for participation by the investigators

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
1-year relapse-free survival rate | 1-year period after randomization
  The rate of no relapse within 1 year

SECONDARY OUTCOMES:
Time to relapse (days) | 1-year period after administration of rituximab therapy
  Number of days from randomization to occurrence of first relapse
Proportion of patients with a relapse | 6 months period after administration of rituximab therapy
  The proportion of patients with relapse
B-Cell Recovery Time | 1-year period after administration of rituximab therapy
  Time to the first detection of CD19+ cells above 1% of total CD45+ lymphocytes after CD19+ cell depletion
The effect of rituximab on peripheral blood B cell subsets and T cell subsets to highlight biomarkers useful for monitoring response to rituximab treatment. | 1-year period after administration of rituximab therapy
  Using fluorescence-activated cell sorting (FACS), peripheral blood B cell subsets and T cell subsets will be measured as at baseline, before and after infusion of rituximab at 3,6,12 months, and when relapse.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1-year period after administration of rituximab therapy
  It is a binary variable (1/0). The variable would be setted as "1" if any adverse events occurs including infusion-related reactions, infection (upper respiratory tract infection, hepatitis B virus reactivation, herpes zoster infection, pneumocystis pneumonia, etc), persistent hypogammaglobulinaemia, encephalopathy, severe neutropenia, fatal pulmonary fibrosis, ulcerative colitis, Crohn's disease and fulminant myocarditis etc. Adverse events will be graded according to the Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Children's Hospital Affiliated to Zhengzhou University/Henan Children's Hospital, Zhengzhou, Henan
  - Wuhan Children's Hospital,Tongji Medical College, Huazhong University of Science and Technology., Wuhan, Hubei
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Zhongshan University, Guanzhou
  - Shandong Provincial Hospital Affiliated to Shandong University, Shandong
  - Children's Hospital of Fudan University, Shanghai
  - Xuzhou Children's Hospital, Xuzhou

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to researchers with a clear research plan and hypothesis, with the appropriate team in place to undertake the work.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When the article has been published with no end date
Access Criteria: Requests for access to data from the RTXFIRPedINS trial should be addressed to the corresponding author at hxu@shmu.edu.cn. The individual participant data collected during the trial (including the data dictionary) will be available, after de-identification. All proposals requesting data access will need to have a research plan and specify how the data will be used, and all proposals will need the approval of the trial coinvestigator team (or individual(s) subsequently delegated this responsibility) before data release.

REFERENCES:
- [Derived] Liu J, Shen Q, Xie L, Wang J, Li Y, Chen J, Fang X, Tang X, Qian B, Xu H. Protocol for an open-label, single-arm, multicentre clinical study to evaluate the efficacy and safety of rituximab in the first episode of paediatric idiopathic nephrotic syndrome. BMJ Open. 2022 Oct 12;12(10):e064216. doi: 10.1136/bmjopen-2022-064216. PMID 36223961

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT04783675/SAP_000.pdf